CLINICAL TRIAL: NCT02290808
Title: First-time Parents Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Lead Investigator, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 133614
Record Dates: First submitted 2014-04-19; First posted 2014-11-14 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Physical Activity
Keywords: physical; activity; exercise; new-parents; intervention; theory-based
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theory-based group (Experimental): The theory-based intervention group will receive strategies based on the Theory of Planned Behaviour to help increase physical activity among couples. Parents will receive materials on how to work together.
  Interventions: Behavioral: Theory-based group
- Information group (No Intervention): The information group will serve as the control group and will receive informational materials on the benefits of physical activity.

INTERVENTIONS:
Behavioral: Theory-based group — Workbooks and mini-counselling sessions will be provided to participants in this group.
  Arms: Theory-based group

SUMMARY:
This study will be investigating whether a theory-based physical activity intervention can maintain/improve moderate to vigorous intensity physical activity measured via accelerometry of new parents over the eight months of having a child compared to a control group of new parents.

Hypothesis: The theory-based condition will change salient underlying motives (theory of planned behaviour constructs) for physical activity. Health-related fitness and quality of life will also be higher for this condition in comparison to the control condition. (Note: improvements in both groups of mothers may occur due to recovery from pregnancy, but our hypotheses will still hold). All outcomes will remain significantly higher at eight months in the theory-based condition compared to the standard condition

DETAILED DESCRIPTION:
Clearly the prevention of chronic disease through physical activity promotion is an important research area. Identifying critical life transitions in people's physical activity behaviours may illuminate the most opportune intervention apertures for chronic disease prevention. A substantive evidence base now indicates that parenthood is one of these critical transition points for physical activity decline. Our proposed study will examine whether a brief, theory-based, and cost-effective intervention can help maintain/improve the physical activity behaviours of new parents in their first eight months of the parenthood experience. The study represents the first couple-based physical activity initiative in the parenthood literature; prior research has only focused on mothers and has shown short-term changes in physical activity that return to baseline levels after approximately one month. In light of the potential for couples to provide important sources of social support for the other parent within the household, it would seem remiss not to consider parenting interventions that are directed and evaluated at the dyadic level. Furthermore, couple-based interventions in other populations and other health behaviour domains have been shown as more effective than individual-level intervention. The long-term impact of this study, if the results support our hypotheses, has utility to prevent or curb the decline of physical activity habits based on our findings. This research has the clear potential to be applied to population-level knowledge translation sources such as prenatal classes, physician offices, and other early parent learning/counselling avenues.

Parents will be measured at baseline (2 months post partum) with two assessment points at six weeks (3.5 months post partum) and three months (5 months post partum) and a final follow-up assessment six months later (8 months post partum). The content of the theory-based intervention was derived from the results of our prior CDA and SSHRC-funded longitudinal trial of new parents using the theory of planned behaviour to predict changes in physical activity, the content used in prior pilot-level studies that has already been successful in changing short-term physical activity in mothers 26-30, and the content of our current CIHR-funded study of physical activity goal planning.

Primary Research Question

1) Does the theory-based condition improve adherence to regular physical activity among new parents when compared to those in the control condition at eight months after the birth of their first child? Hypothesis: Adherence will be higher for parents in the theory-based condition in comparison to parents in the control condition after controlling for possible confounds. The adherence effect may wane over time from the initial measurement period of two months after the onset of parenthood but all outcomes will remain significantly higher at eight months.

Secondary Research Questions

1. Does the theory-based condition improve motivational, health-related quality of life, and health-related fitness outcomes among new parents when compared to those in the control condition at eight months after the onset of parenthood? Hypothesis: The theory-based condition will change salient underlying motives (theory of planned behaviour constructs) for physical activity because its basis is from the key results of our prior longitudinal trial of new parents. Health-related fitness and quality of life, will also be higher for this condition in comparison to the control condition, (footnote: improvements in both groups of mothers may occur due to recovery from pregnancy, but our hypotheses will still hold). All outcomes will remain significantly higher at eight months in the theory-based condition compared to the standard physical activity education group.
2. Can group differences among new parents with regard to these motivational, behavioural, and health-related fitness outcomes be explained through a mediation model?

   Hypothesis: The covariance of the assigned conditions (theory-based, standard) on adherence will be explained by changes in the salient underlying motives for physical activity (i.e., manipulation check). In turn, the covariance between these salient underlying motives and health-related outcomes will be explained by physical activity adherence among conditions.
3. Can motivational variables predict adherence? Do these differ by condition?

   Hypothesis: The approach will test Ajzen's 39 theory of planned behavior. Affective attitude and perceived behavioural control will predict intention, intention will predict adherence across conditions similar to our prior study with this population 41.
4. Is there a seasonal, initial physical activity status, mental health or gender difference across primary outcomes by assigned condition?

Hypothesis: No differences in gender or season are hypothesized based on our lack of evidence in the prior trial41, but these are exploratory research questions because there is limited research at present to make any definitive statement. The examination of whether the intervention affects maintenance or increases in baseline physical activity via stratification of baseline values will also be explored as will the assessment of baseline depression and anxiety.

Recruitment: We began feasibility recruitment and procedures last year in order to establish our protocol, and pilot our intervention material. Based on this feasibility study, participant recruitment is being achieved with both active (pregnancy class visits) and passive recruitment techniques (notice of research and poster). The active recruitment is being conducted through community organizations offering prenatal classes and programming for first-time parents. The project coordinator and research assistants associated with this project are the main point of contact for potential participants. Organizations are contacted by the research coordinator and asked if they are interested in giving 10 minutes of time (prenatal class, workshop).

ELIGIBILITY:
Inclusion Criteria:

* Married or common law couples
* Living in Greater Victoria
* Expecting first child
* 18 years of age or older

Exclusion Criteria:

* younger than 18
* Expecting second or third child

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change in Objective and Self-report Physical activity | Baseline, 6 weeks, 3.5 months, and 6 months
  Physical activity will be measured objectively for 7 consecutive days using the wGT3X-BT Activity Monitor combined with self-report of PA using the Godin Leisure-Time Exercise Questionnaire (LSI) at each time period.

SECONDARY OUTCOMES:
Demographic information | Baseline
  Basic information on gender, age, ethnicity, income, education level will be gathered.
Health measures | Baseline and 6 months
  Information on leave status, child care status, diet, sleep (Pittsburgh sleep quality index) and breastfeeding status, smoking, alcohol consumption will be included in this assessment.
Motivation for physical activity | Baseline, 6 weeks, 3.5 months, 6 months
  Motivation will be measured using the constructs of the theory of planned behaviour. Items will measure all components of the model (affective attitude, instrumental attitude, injunctive norm, descriptive norm, perceived control, planning) including behavioural, normative, and control beliefs.
Health related quality of life/psychosocial distress | Baseline, 6 weeks, 3.5 months, 6 months
  This will be assessed with parents using the Satisfaction with Life Scale. In addition, we will assess depressive and anxiety symptoms with the Hospital Anxiety and Depression Scale (HADS), which also has sound reliability and validity compared to similar instruments.
Health related fitness | Baseline and 6 months
  We will assess the key components of health-related physical fitness including body composition, aerobic fitness and musculoskeletal fitness which are valid for males and females.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD., Principal Investigator — University of Victoria; Mark Beauchamp, PhD, Study Director — University of British Columbia; Chris Blanchard, PhD, Study Director — Dalhousie; Darren Warburton, PhD, Study Director — University of British Columbia; Danielle Downs, PhD, Study Director — Penn State University
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

REFERENCES:
- [Background] Warburton DE, Charlesworth S, Ivey A, Nettlefold L, Bredin SS. A systematic review of the evidence for Canada's Physical Activity Guidelines for Adults. Int J Behav Nutr Phys Act. 2010 May 11;7:39. doi: 10.1186/1479-5868-7-39. PMID 20459783
- [Background] Warburton DE, Nicol CW, Bredin SS. Health benefits of physical activity: the evidence. CMAJ. 2006 Mar 14;174(6):801-9. doi: 10.1503/cmaj.051351. PMID 16534088
- [Background] Warburton DE, Nicol CW, Bredin SS. Prescribing exercise as preventive therapy. CMAJ. 2006 Mar 28;174(7):961-74. doi: 10.1503/cmaj.1040750. PMID 16567757
- [Background] Warburton DE, Katzmarzyk PT, Rhodes RE, Shephard RJ. Evidence-informed physical activity guidelines for Canadian adults. Can J Public Health. 2007;98 Suppl 2:S16-68. PMID 18213940
- [Background] Colley RC, Garriguet D, Janssen I, Craig CL, Clarke J, Tremblay MS. Physical activity of Canadian children and youth: accelerometer results from the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2011 Mar;22(1):15-23. PMID 21510586
- [Background] Colley RC, Garriguet D, Janssen I, Craig CL, Clarke J, Tremblay MS. Physical activity of Canadian adults: accelerometer results from the 2007 to 2009 Canadian Health Measures Survey. Health Rep. 2011 Mar;22(1):7-14. PMID 21510585
- [Background] Bellows-Riecken KH, Rhodes RE. A birth of inactivity? A review of physical activity and parenthood. Prev Med. 2008 Feb;46(2):99-110. doi: 10.1016/j.ypmed.2007.08.003. Epub 2007 Aug 15. PMID 17919713
- [Background] Craig CL, Russell SJ, Cameron C, Bauman A. Twenty-year trends in physical activity among Canadian adults. Can J Public Health. 2004 Jan-Feb;95(1):59-63. doi: 10.1007/BF03403636. PMID 14768744
- [Background] Craig S, Goldberg J, Dietz WH. Psychosocial correlates of physical activity among fifth and eighth graders. Prev Med. 1996 Sep-Oct;25(5):506-13. doi: 10.1006/pmed.1996.0083. PMID 8888317
- [Background] Walker LO. Weight gain after childbirth: a women's health concern? Ann Behav Med. 1995 Spring;17(2):132-41. doi: 10.1007/BF02895062. PMID 18425664
- [Background] Walker LO. Weight-related distress in the early months after childbirth. West J Nurs Res. 1998 Feb;20(1):30-44. doi: 10.1177/019394599802000103. PMID 9473966
- [Background] Downs DS, Hausenblas HA. Exercising for two: examining pregnant women's second trimester exercise intention and behavior using the framework of the theory of planned behavior. Womens Health Issues. 2003 Nov-Dec;13(6):222-8. PMID 14675791
- [Background] Hausenblas H, Downs DS, Giacobbi P, Tuccitto D, Cook B. A multilevel examination of exercise intention and behavior during pregnancy. Soc Sci Med. 2008 Jun;66(12):2555-61. doi: 10.1016/j.socscimed.2008.02.002. Epub 2008 Mar 26. PMID 18372085
- [Background] Rhodes RE, Blanchard CM, Benoit C, Levy-Milne R, Naylor PJ, Symons Downs D, Warburton DE. Physical activity and sedentary behavior across 12 months in cohort samples of couples without children, expecting their first child, and expecting their second child. J Behav Med. 2014 Jun;37(3):533-42. doi: 10.1007/s10865-013-9508-7. Epub 2013 Apr 19. PMID 23606310
- [Background] Rhodes RE, Blanchard CM, Benoit C, Levy-Milne R, Naylor PJ, Symons Downs D, Warburton DE. Social cognitive correlates of physical activity across 12 months in cohort samples of couples without children, expecting their first child, and expecting their second child. Health Psychol. 2014 Aug;33(8):792-802. doi: 10.1037/a0033755. Epub 2013 Aug 5. PMID 23914818
- [Background] McIntyre CA, Rhodes RE. Correlates of leisure-time physical activity during transitions to motherhood. Women Health. 2009 Jan-Feb;49(1):66-83. doi: 10.1080/03630240802690853. PMID 19485235
- [Background] Mailey EL, McAuley E. Impact of a brief intervention on physical activity and social cognitive determinants among working mothers: a randomized trial. J Behav Med. 2014 Apr;37(2):343-55. doi: 10.1007/s10865-013-9492-y. Epub 2013 Jan 22. PMID 23338616
- [Background] Cramp AG, Brawley LR. Moms in motion: a group-mediated cognitive-behavioral physical activity intervention. Int J Behav Nutr Phys Act. 2006 Aug 22;3:23. doi: 10.1186/1479-5868-3-23. PMID 16925809
- [Background] Fahrenwald NL, Atwood JR, Walker SN, Johnson DR, Berg K. A randomized pilot test of "Moms on the Move": a physical activity intervention for WIC mothers. Ann Behav Med. 2004 Apr;27(2):82-90. doi: 10.1207/s15324796abm2702_2. PMID 15026292
- [Background] Miller YD, Trost SG, Brown WJ. Mediators of physical activity behavior change among women with young children. Am J Prev Med. 2002 Aug;23(2 Suppl):98-103. doi: 10.1016/s0749-3797(02)00484-1. PMID 12133744
- [Background] Fjeldsoe BS, Miller YD, Marshall AL. MobileMums: a randomized controlled trial of an SMS-based physical activity intervention. Ann Behav Med. 2010 May;39(2):101-11. doi: 10.1007/s12160-010-9170-z. PMID 20174902
- [Background] Burke V, Giangiulio N, Gillam HF, Beilin LJ, Houghton S. Physical activity and nutrition programs for couples: a randomized controlled trial. J Clin Epidemiol. 2003 May;56(5):421-32. doi: 10.1016/s0895-4356(02)00610-8. PMID 12812815
- [Background] Black DR, Gleser LJ, Kooyers KJ. A meta-analytic evaluation of couples weight-loss programs. Health Psychol. 1990;9(3):330-47. doi: 10.1037//0278-6133.9.3.330. PMID 2140323
- [Background] Burke V, Giangiulio N, Gillam HF, Beilin LJ, Houghton S, Milligan RA. Health promotion in couples adapting to a shared lifestyle. Health Educ Res. 1999 Apr;14(2):269-88. doi: 10.1093/her/14.2.269. PMID 10387506
- [Background] Dzator JA, Hendrie D, Burke V, Gianguilio N, Gillam HF, Beilin LJ, Houghton S. A randomized trial of interactive group sessions achieved greater improvements in nutrition and physical activity at a tiny increase in cost. J Clin Epidemiol. 2004 Jun;57(6):610-9. doi: 10.1016/j.jclinepi.2003.10.009. PMID 15246129
- [Background] Baranowski T, Anderson C, Carmack C. Mediating variable framework in physical activity interventions. How are we doing? How might we do better? Am J Prev Med. 1998 Nov;15(4):266-97. doi: 10.1016/s0749-3797(98)00080-4. PMID 9838973
- [Background] Rhodes RE, Pfaeffli LA. Mediators of physical activity behaviour change among adult non-clinical populations: a review update. Int J Behav Nutr Phys Act. 2010 May 11;7:37. doi: 10.1186/1479-5868-7-37. PMID 20459781
- [Background] Hamilton K, White KM. Identifying key belief-based targets for promoting regular physical activity among mothers and fathers with young children. J Sci Med Sport. 2011 Mar;14(2):135-42. doi: 10.1016/j.jsams.2010.07.004. Epub 2010 Aug 30. PMID 20800540
- [Background] Rhodes RE, Naylor PJ, McKay HA. Pilot study of a family physical activity planning intervention among parents and their children. J Behav Med. 2010 Apr;33(2):91-100. doi: 10.1007/s10865-009-9237-0. Epub 2009 Nov 24. PMID 19937106
- [Background] Rhodes RE, Murray H, Temple VA, Tuokko H, Higgins JW. Pilot study of a dog walking randomized intervention: effects of a focus on canine exercise. Prev Med. 2012 May;54(5):309-12. doi: 10.1016/j.ypmed.2012.02.014. Epub 2012 Mar 1. PMID 22405707
- [Background] Gainforth HL, Berry T, Faulkner G, Rhodes RE, Spence JC, Tremblay MS, Latimer-Cheung AE. Evaluating the uptake of Canada's new physical activity and sedentary behavior guidelines on service organizations' websites. Transl Behav Med. 2013 Jun;3(2):172-9. doi: 10.1007/s13142-012-0190-z. PMID 24073168
- [Background] Charlesworth S, Foulds HJ, Burr JF, Bredin SS. Evidence-based risk assessment and recommendations for physical activity clearance: pregnancy. Appl Physiol Nutr Metab. 2011 Jul;36 Suppl 1:S33-48. doi: 10.1139/h11-061. PMID 21800947
- [Background] Rhodes RE, Temple VA, Tuokko HA. Evidence-based risk assessment and recommendations for physical activity clearance: cognitive and psychological conditions. Appl Physiol Nutr Metab. 2011 Jul;36 Suppl 1:S113-53. doi: 10.1139/h11-041. PMID 21800939
- [Background] Atkins DC. Using multilevel models to analyze couple and family treatment data: basic and advanced issues. J Fam Psychol. 2005 Mar;19(1):98-110. doi: 10.1037/0893-3200.19.1.98. PMID 15796656
- [Background] King AC, Stokols D, Talen E, Brassington GS, Killingsworth R. Theoretical approaches to the promotion of physical activity: forging a transdisciplinary paradigm. Am J Prev Med. 2002 Aug;23(2 Suppl):15-25. doi: 10.1016/s0749-3797(02)00470-1. PMID 12133734
- [Background] Travers KD. The social organization of nutritional inequities. Soc Sci Med. 1996 Aug;43(4):543-53. doi: 10.1016/0277-9536(95)00436-x. PMID 8844955
- [Background] Dumas JE, Lynch AM, Laughlin JE, Phillips Smith E, Prinz RJ. Promoting intervention fidelity. Conceptual issues, methods, and preliminary results from the EARLY ALLIANCE prevention trial. Am J Prev Med. 2001 Jan;20(1 Suppl):38-47. doi: 10.1016/s0749-3797(00)00272-5. PMID 11146259
- [Background] Webb TL, Sheeran P. Mechanisms of implementation intention effects: the role of goal intentions, self-efficacy, and accessibility of plan components. Br J Soc Psychol. 2008 Sep;47(Pt 3):373-95. doi: 10.1348/014466607X267010. Epub 2007 Dec 18. PMID 18096108
- [Background] Brown SG, Rhodes RE. Relationships among dog ownership and leisure-time walking in Western Canadian adults. Am J Prev Med. 2006 Feb;30(2):131-6. doi: 10.1016/j.amepre.2005.10.007. PMID 16459211
- [Background] Rhodes RE, Plotnikoff RC. Can current physical activity act as a reasonable proxy measure of future physical activity? Evaluating cross-sectional and passive prospective designs with the use of social cognition models. Prev Med. 2005 May;40(5):547-55. doi: 10.1016/j.ypmed.2004.07.016. PMID 15749137
- [Background] Rhodes RE, Warburton DE, Bredin SS. Predicting the effect of interactive video bikes on exercise adherence: An efficacy trial. Psychol Health Med. 2009 Dec;14(6):631-40. doi: 10.1080/13548500903281088. PMID 20183536
- [Background] Casiro NS, Rhodes RE, Naylor PJ, McKay HA. Correlates of intergenerational and personal physical activity of parents. Am J Health Behav. 2011 Jan-Feb;35(1):81-91. doi: 10.5993/ajhb.35.1.8. PMID 20950161
- [Background] Janz KF. Validation of the CSA accelerometer for assessing children's physical activity. Med Sci Sports Exerc. 1994 Mar;26(3):369-75. PMID 8183103
- [Background] Strath SJ, Brage S, Ekelund U. Integration of physiological and accelerometer data to improve physical activity assessment. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S563-71. doi: 10.1249/01.mss.0000185650.68232.3f. PMID 16294119
- [Background] Welk GJ. Principles of design and analyses for the calibration of accelerometry-based activity monitors. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S501-11. doi: 10.1249/01.mss.0000185660.38335.de. PMID 16294113
- [Background] Godin G, Jobin J, Bouillon J. Assessment of leisure time exercise behavior by self-report: a concurrent validity study. Can J Public Health. 1986 Sep-Oct;77(5):359-62. No abstract available. PMID 3791117
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Jacobs DR Jr, Ainsworth BE, Hartman TJ, Leon AS. A simultaneous evaluation of 10 commonly used physical activity questionnaires. Med Sci Sports Exerc. 1993 Jan;25(1):81-91. doi: 10.1249/00005768-199301000-00012. PMID 8423759
- [Background] Lee RG, Garvin T. Moving from information transfer to information exchange in health and health care. Soc Sci Med. 2003 Feb;56(3):449-64. doi: 10.1016/s0277-9536(02)00045-x. PMID 12570966
- [Derived] Rhodes RE, Blanchard CM, Hartson KR, Symons Downs D, Warburton DER, Beauchamp MR. Affective Response to Exercise and Affective Judgments as Predictors of Physical Activity Intention and Behavior among New Mothers in their first 6-Months Postpartum. Ann Behav Med. 2023 Apr 12;57(4):344-353. doi: 10.1093/abm/kaac067. PMID 36745018
- [Derived] Rhodes RE, Blanchard CM, Quinlan A, Symons Downs D, Warburton DER, Beauchamp MR. Couple-Based Physical Activity Planning for New Parents: A Randomized Trial. Am J Prev Med. 2021 Oct;61(4):518-528. doi: 10.1016/j.amepre.2021.04.020. Epub 2021 Jul 3. PMID 34226094
- [Derived] Quinlan A, Rhodes RE, Beauchamp MR, Symons Downs D, Warburton DER, Blanchard CM. Evaluation of a physical activity intervention for new parents: protocol paper for a randomized trial. BMC Public Health. 2017 Nov 9;17(1):875. doi: 10.1186/s12889-017-4874-7. PMID 29121884